CLINICAL TRIAL: NCT00109499
Title: An Open-label, Phase I, Single Administration, Dose- Escalation Study of AdGVPEDF.11D in Neovascular Age-related Macular Degeneration (AMD)
Brief Title: Study of AdGVPEDF.11D in Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Masking: None | Purpose: Treatment
Other Study IDs: GV-003.001
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Macular Degeneration
Keywords: Wet Age-Related Macular Degeneration; Age-Related Maculopathies
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Drug: AdGVPEDF.11D

SUMMARY:
The primary purpose of this study is to assess the safety of AdGVPEDF.11D when given to patients with "wet" age-related macular degeneration (AMD). AdGVPEDF.11D is a replication deficient (E1, E3 and E4 deleted) adenovirus vector containing the gene for the PEDF (pigment epithelium-derived factor) protein. PEDF is a protein that naturally exists in the human eye, but whose levels are altered in diseases characterized by ocular neovascularization like AMD. The PEDF protein is known to have anti-angiogenic effects or, in other words, it has the ability to inhibit growth of new blood vessels.

AdGVPEDF.11D will be delivered once via intravitreal injection into one eye. The injected eye will be the eye with the worst visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years;
* Severe neovascular AMD in at least one eye responsible for a best corrected vision of 20/200 or worse in the study eye (if both eyes have neovascular AMD and equal visual acuity scores, the study eye will be determined by the investigator);
* Best corrected visual acuity in the fellow eye must be equal to or better than the study eye;
* Fluorescein angiography of the study eye must show evidence of a leaking subfoveal choroidal neovascular lesion. The subfoveal component must consist of CNV (choroidal neovascularization), blood or fibrosis. The total size of the lesion must be ≤12 MPS disc areas. The presence of a leaking subfoveal choroidal neovascular lesion will be evaluated by the investigator at the clinical site to determine patients' eligibility.
* Must not be candidates for (including patients who have had treatment with either modality in the past and are no longer candidates) or must have refused treatment with subfoveal laser photocoagulation or PDT (photodynamic therapy);
* Informed consent;
* Able to comply with protocol requirements including follow-up visits.

Exclusion Criteria:

* Liver enzymes > 2 x ULN (ALT, AST, bilirubin);
* Clinical evidence of active infection of any type, including adenovirus, hepatitis A, B, or C virus or HIV virus;
* Other treatment for AMD in the study eye within the last twelve weeks prior to Day 1;
* Other experimental medications within the last four weeks prior to Day 1;
* Significant retinal disease other than neovascular AMD, such as diabetic retinopathy or retinal vascular occlusion;
* Significant non-retinal disease such as ocular atrophy;
* Cataract or other significant media opacity that might compromise examination and photography of the posterior segment;
* Other causes of choroidal neovascularization such as pathologic myopia ( > 8 diopters), ocular histoplasmosis or angioid streaks;
* Evidence of inflammation (grade 1 or higher) in the anterior and/or posterior chambers;
* Cataract surgery or submacular surgery within 3 months;
* Prior ocular treatment with radiation;
* Known allergy to fluorescein;
* Abnormal prothrombin or partial thromboplastin time ( > 1.5 X ULN) or anticoagulant therapy that cannot be withheld for treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Transplantation Laboratory, Los Angeles, California
  - UCLA - Jules Stein Eye Research Center, Los Angeles, California
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Johns Hopkins Hospital School of Medicine, Baltimore, Maryland
  - Kresge Eye Institute, Detroit, Michigan
  - Casey Eye Institute, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington